CLINICAL TRIAL: NCT04697589
Title: Acute Dose-response Effect of a Proprietary Botanical Blend Rich in Polyphenols on Flow-mediated Dilation in Healthy Subjects: Randomized, Cross-over, Double-blind Clinical Study
Brief Title: Acute Effect of a Proprietary Botanical Blend Rich in Polyphenols on Flow-mediated Dilation in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Activ'inside (Industry)
Collaborators: CIC Inserm 1405, University Hospital Clermont-Ferrand, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: FMD1-AI-2020
Record Dates: First submitted 2021-01-05; First posted 2021-01-06 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: endothelial function; healthy adults; grape and blueberry extracts; flavanol monomers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SBRP 300 mg (Experimental): 300 mg standardized botanical blend rich in polyphenols (SBRP) and especially in monomers of flavanols.
  Interventions: Dietary Supplement: Memophenol 300 mg
- SBRP 600 mg (Experimental): 600 mg standardized botanical blend rich in polyphenols (SBRP) and especially in monomers of flavanols.
  Interventions: Dietary Supplement: Memophenol 600 mg
- Placebo (Placebo Comparator): Colored maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Memophenol 300 mg — 300 mg a proprietary, standardized botanical blend rich in polyphenols (SBRP) and especially in monomers of flavanols.
  Arms: SBRP 300 mg
Dietary Supplement: Memophenol 600 mg — 600 mg a proprietary, standardized botanical blend rich in polyphenols (SBRP) and especially in monomers of flavanols.
  Arms: SBRP 600 mg
Dietary Supplement: Placebo — Colored maltodextrin
  Arms: Placebo

SUMMARY:
It is well established that endothelial dysfunction is an early predictor of cardiovascular events in at-risk patients. Finding safe and effective product able to improve endothelial function is of public health interest.

Many clinical studies have shown that monomer of flavanols from cocoa significantly improved endothelial function, in particular endothelium-dependent flow-mediated dilation (ED-FMD) after a single dose. Grape is also a main source of flavanol monomers, that's why many human studies have shown significant effects of grape-derived products on endothelial function within 2 hours following a single dose intake.

The objective of this study is to assess the effect of 2 doses of a proprietary and standardised botanical blend rich in polyphenols (SBRP), on ED-FMD in fasting conditions, in comparison to a placebo, in healthy adults. This blend is made of two botanical extracts: a grape extract and a blueberry extract. In order to provide supportive evidence on the mechanisms and biological plausibility to the clinical effects of the product, appropriate biological parameters and circulating metabolites will be assayed.

ELIGIBILITY:
Inclusion Criteria:

* Presenting at least two of the following risks of suboptimal endothelial function (but not under prescribed drug for this reason):
* Overweight, defined by: 25 ≤ BMI < 30 kg/m2;
* Central obesity defined according to IDE criteria (2009): for European subjects, waist circumference ≥ 94 cm (with a tolerance of -10%);
* High Normal Blood pressure defined according to ESC/ESH guidelines (2013): Systolic Blood Pressure ≥ 130 and ≤ 139 mmHg or Diastolic Blood Pressure ≥ 85 and ≤ 89 mmHg;
* Considered healthy based on their self-declaration and physical examination;
* Subjects capable of and willing to comply with the protocol and to give their written informed consent.
* Subjects affiliated with a social security scheme.

Non-inclusion Criteria:

* Metabolic abnormality or major cardiovascular risk factor, such as (but not limited to):
* clinically significant arrhythmia,
* diabetes mellitus (type I or II),
* chronic kidney disease.
* Consumption of food supplement(s) currently or within the past 4 weeks before entry into the study, such as but not limited to: botanicals, vitamins, minerals, amino acids;
* Smoking > 5 cigarettes/ day and > 5 pack-years for at least 2 years;
* Use of any type of medication currently or within 2 months before entry into the study (more especially antihypertensive drug);
* Use of any narcotic drug (including cannabis) within 2 months before entry into the study detected by the self-declaration of the participant and/ or by the urine THC test ;
* Endurance sport activities > 5 h/ week;
* Self-reported alcohol intake >10 units/ week (1 unit = 1 standard glass)
* Weight change > 5% of total body weight within the 3 months before V1;
* Currently under prescribed diet regimen, whatever the reason;
* Any intolerance or allergy documented or suspected to one of the components of the study products or to the Glyceryl trinitrate (GTN);
* Any contraindication to the GTN drug:
* severe hypotension,
* obstructive cardiomyopathy,
* myocardial infarction,
* intracranial hypertension,
* sildenafil intake (occasionally or regularly). .
* Subject presenting a psychological or linguistic inability to sign the informed consent;
* Subject under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision;
* Subject participating in another biomedical study or participation in another study within the 3 months before entry into this study;
* Any regulatory reason according to national applicable regulation.

Exclusion criteria :

Volunteers whose fasting blood sample at V0 will reveal a pathological level of glycaemia (> 1,26 g/L) and/ or a dyslipidemia (example : triacylglycerol > 1,75 g/L) will be excluded.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Change in endothelium-dependent flow-mediated dilation (ED-FMD) | Between Baseline (Before product intake) and 2 hours after product intake
  ED-FMD : maximal change in the diameter of the brachial artery induced by increased flow, expressed in percentage (%) of the basal diameter.

SECONDARY OUTCOMES:
Change in endothelium-independent vasodilation (EIVD) | Between Baseline (Before product intake) and 2 hours after product intake
  EIVD : Baseline diameter of the brachial artery will be assessed, and the increase in diameter of the brachial artery after application of glyceryl trinitrate will be measured .
Change in diastolic blood pressure | Between Baseline (Before product intake) and 2 hours after product intake
  Blood pressure will be measured 3 times separated by 3-minute intervals. The average of the 3 measurements will be calculated.
Change in systolic blood pressure | Between Baseline (Before product intake) and 2 hours after product intake
  Blood pressure will be measured 3 times separated by 3-minute intervals. The average of the 3 measurements will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle Pickering, Principal Investigator — CIC Inserm 1405, University Hospital Clermont-Ferrand, France
Locations (1):
- CIC Inserm 1405, University Hospital Clermont-Ferrand,, Clermont-Ferrand, France